CLINICAL TRIAL: NCT06644677
Title: Development of a Third-Generation Nanopore HPV Integration Site Detection Kit for Precise Prediction of Cervical Cancer Prognosis
Brief Title: Third-Generation Nanopore HPV Integration Site for Precise Prediction of Cervical Cancer Prognosis
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhang Fuquan, Professor, Peking Union Medical College Hospital
Other Study IDs: CHINTIGER
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2019-09

CONDITIONS: Cervical Cancers; HPV Testing; Nanopore Sequencing; HPV Integration Site Detection; Rapid Diagnosis
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — the patient's cells, extracted DNA, or RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Advanced-stage cervical cancer patients group (Stage IIIB and beyond)
  Interventions: Diagnostic Test: HPV integration

INTERVENTIONS:
Diagnostic Test: HPV integration — Collect late-stage cervical cancer (Stage IIIB and beyond) and post-treatment recurrence and metastasis specimens (TCT, tissue) associated with HPV infection. Utilize third-generation nanopore technology to detect the integration sites of HPV DNA based on the principle of probe hybridization capture. Obtain information on HPV integration and hot spot genes in the samples. By analyzing the integration of HPV in primary and recurrent/metastatic tissues, identify insertions and gene alterations associated with recurrence/metastasis, and develop a predictive formula.

SUMMARY:
Cervical cancer is a significant health threat to women, with over 500,000 new cases and approximately 342,000 deaths worldwide annually, and about 107,000 new cases in China with 51,000 fatalities. Current screening methods include HPV testing, cytology, colposcopy, and biopsy, but none can detect HPV genome integration in persistently positive patients.

Our team has analyzed over 200 cervical cell samples using third-generation nanopore technology, focusing on HPV integration sites. We've developed a proprietary long-fragment capture and sequencing method (reads averaging 2-5kb) that identifies precise HPV insertion points and detects the complete Human-Virus-Human (H-V-H) viral insertion sequence. We found overlaps in HPV integration genes across different stages of cervical intraepithelial neoplasia (CIN) and in cancer patients with recurrence and metastasis, suggesting potential biomarkers for tumor progression and poor prognosis.

We also analyzed HPV sequence proportions and gene insertion numbers in samples from patients before and after radical radiochemotherapy, providing insights into treatment efficacy and prognosis. Our study aims to use a domestic nanopore sequencing platform and probes tailored to Chinese HPV infection patterns to detect integration sites in late-stage cervical cancer and post-treatment recurrence/metastasis patients. We aim to optimize our method to complete the entire detection process within eight hours, expanding the technology's application in point-of-care diagnostics and decentralization.

DETAILED DESCRIPTION:
Cervical cancer is the most common malignant tumor of the reproductive tract, posing a serious threat to women's health. According to data from the World Health Organization (WHO), there are over 500,000 new cases of cervical cancer globally each year, with approximately 342,000 deaths. In China, there are about 107,000 new cases annually, with around 51,000 patients dying from cervical cancer. The market for detection is vast and continues to grow. The main methods of examination after cervical cancer screening and treatment include HPV testing, cytological screening, colposcopy, and cervical biopsy. All HPV tests on the market are qualitative and semi-quantitative, and there is currently no product on the market that can detect whether HPV integrates into the genome in patients with persistent HPV positivity.

Our team, in previous research, enrolled over 200 cervical cell samples, including those from patients with high-risk HPV infection without intraepithelial neoplasia, cervical intraepithelial neoplasia (CIN) I, CIN II, CIN III, and samples from locally advanced cervical cancer before and after radiochemotherapy at multiple time points. Using third-generation nanopore technology, we have completed experiments and analysis on 93 cervical cell samples. Based on the probe hybridization capture principle, we enriched and sequenced the integration sites of HPV viral DNA. Preliminary conclusions are as follows:

1. Through our self-developed experimental technology process, we achieved long-fragment virus capture and sequencing (average read length 2-5kb), identifying HPV insertion sites and more precise genomic localization. Moreover, nanopore long-fragment sequencing can detect the complete Human-Virus-Human (H-V-H) viral insertion structure sequence.
2. There is a certain proportion of overlap between the HPV insertion genes in the inflammation group, CIN I, CIN II, CIN III groups, and the HPV insertion genes in cancer patients with recurrence and metastasis, which can further assist in screening for molecular markers related to tumor progression and poor prognosis.
3. The proportion of HPV sequences and the number of inserted genes in patient samples before and after radical radiochemotherapy can further assess the effectiveness of treatment and prognosis, providing support data for pre-treatment intervention and risk warning.

The goal of this study is to collaborate with a domestically produced nanopore sequencing platform and self-designed probes targeting the characteristics of HPV infection in the Chinese population. We aim to conduct insertion site detection on cohorts of late-stage cervical cancer (stage IIIB and beyond) and patients with recurrence and metastasis after radical cervical cancer radiochemotherapy. We will further establish and optimize the long-fragment virus enrichment method and nanopore sequencing experimental process to complete the entire detection process within one working day (8 hours). This will also expand the application of the technology in bedside diagnosis and decentralized directions.

ELIGIBILITY:
Inclusion Criteria:

* A. Undergoing radical radiochemotherapy at our institution or a collaborating institution; B. Pathologically confirmed as cervical cancer; C. Diagnosed as an advanced-stage patient (FIGO staging IIIB, IIIC, IVA, IVB), or a patient who has experienced local recurrence or distant metastasis after radical radiochemotherapy; D. Capable of regular follow-up visits; E. The patient or their family can understand the research protocol and are willing to participate in this study, providing written informed consent.

Exclusion Criteria:

* A. Confirmed by pathology as neuroendocrine carcinoma of the cervix; B. Have not undergone standardized radical treatment (for the cohort of stage IIIB and later cervical cancer patients, those who have not undergone standardized radical radiochemotherapy must be excluded. For the cohort of patients who have local recurrence or distant metastasis after radical radiochemotherapy, those who have only had cervical cancer surgery and recurrence, and those who have not undergone standardized radiochemotherapy after cervical cancer surgery must be excluded); C. HPV testing is negative, and there is no clear integration site of HPV in the genome; D. The patient or family members are unable to cooperate with the study or cannot provide written informed consent.

Ages: 75 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients enrolled in the study are those with advanced-stage cervical cancer (Stage IIIB and beyond), with TCT procedures performed by radiation oncologists. During the procedure, sterile physiological cotton balls are used to clean away external cervical secretions. A cytobrush is inserted into the cervical lesion or the squamocolumnar junction within the cervical canal to collect samples, rotated 3-4 times, left in place for several seconds, and then placed into a cell preservation fluid, sealed, and sent for testing. As a therapeutic department, the radiation oncology department is heavily involved in the entire process of diagnosis, treatment, and follow-up for cervical cancer patients. During treatment, patients undergo invasive brachytherapy, which has a higher level of sterility requirements and operational difficulty than TCT procedures, hence they are capable of performing TCT specimen collection.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
  Disease-free survival was defined as the period from the diagnosis of cervical cancer to events that included death or disease progression at local, regional, or distant sites or until the date of the last follow-up.

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival was defined as the period from the diagnosis of cervical cancer to the date of death or last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of the patients